CLINICAL TRIAL: NCT00619541
Title: Phase II Study of Sorafenib (Bay 43-9006) and Infusional 5-Fluorouracil in Advanced Hepatocellular Carcinoma.
Brief Title: Study of Sorafenib and Infusional 5-Fluorouracil in Advanced Hepatocellular Carcinoma (HCC)
Acronym: P2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Trial in Medical Oncology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PISADUE
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Sorafenib; Pisa; Ricci; 5-FU; 5FU; 5 FU; Advanced HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): * 5-FU 3000 mg/sqm 48 hours continuous infusion every 14 days
  * Sorafenib 400 mg bid orally continuously
  * 5-FU will be administered for a maximum of 12 cycles.
  * Sorafenib will be administered from the start of treatment in combination with 5-FU until progression of disease.
  Interventions: Drug: Infusional 5-Fluorouracil; Drug: Sorafenib (Bay 43-9006)

INTERVENTIONS:
Drug: Infusional 5-Fluorouracil — 5-FU 3000 mg/sqm 48 hours continuous infusion every 14 days. 5-FU will be administered for a maximum of 12 cycles.
Drug: Sorafenib (Bay 43-9006) — Sorafenib 400 mg bid orally continuously. Sorafenib will be administered from the start of treatment in combination with 5-FU until progression of disease.

SUMMARY:
The purpose of this study is to use Sorafenib + 5-FU to evaluate activity, efficacy, safety, pharmacodynamics (PD) and pharmacokinetics (PK) in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Numerous chemotherapeutic regimens have been tested for use against hepatocellular carcinoma (HCC). HCC is, however, highly resistant to chemotherapy; doxorubicin and 5- fluorouracil containing regimens, alone or in combinations, results in less than a 20% response, with a median survival of less than 4 months. Furthermore even the objective responses are short-lasting. In a metaanalysis of the published randomized studies on HCC, neither doxorubicin nor any chemotherapeutic agent has been shown to have any survival benefit for HCC patients.

Sorafenib (Bay 43-9006) is a novel signal transduction inhibitor that prevent tumor cell proliferation and angiogenesis through blockade of the Raf/Mek/Erk pathway at the level of Raf Kinase and the receptor tyrosine kinases VEGFR-2 and PDGFR-beta.

Recent preclinical studies have shown the activation of Mek-1/2 and its downstream target MAPK in HCC tumors. In a phase II study 137 patients advanced primary liver cancer with have been treated with Sorafenib administered as a single agent. Investigators reported seven patients with partial responses, five minor responses and 59 with stable disease for at least 4 months. Median overall survival was 9.2 months and median time to progression 4.2 months. This study showed that Sorafenib was well tolerated and side-effects were manageable and reversible.

Rationale

5-Fluorouracil (5-FU) is a widely used agent for patients with unresectable advanced HCC, with objective responses rates around 10%. Compared to bolus administration, infusional 5-FU in metastatic colorectal cancers has demonstrated increased activity with less toxicity.

Sorafenib as single agent in HCC has demonstrated activity in terms of objective responses and promising duration of stable disease.

The combination of Sorafenib and 5-FU was evaluated in a phase I study where the drug is associated with different 5FU based schedules with good toxicity profile and objectives responses in particular in colorectal carcinoma.

Based on these data our purpose is to study infusional 5-FU with Sorafenib to evaluate the activity, efficacy, safety, pharmacokinetics and pharmacodynamics of this combination.

Study design and duration of treatment

5-FU 3000 mg/sqm 48 hours continuous infusion every 14 days Sorafenib 400 mg bid orally continuously 5-FU will be administered for a maximum of 12 cycles. Sorafenib will be administered from the start of treatment in combination with 5-FU until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

Screening must be done within 28 days of study drug administration (laboratory evaluations must be done within 7 days). For inclusion in the study, patients must fulfill all of the following criteria:

* Age 18 years.
* Patients should have proven primary HCC according to one of the following criteria:

  * Histological evidence of HCC on a biopsy specimen. Patients with the fibrolamellar subset are excluded, as are any patients with a mixed histology.
  * Cytological evidence of HCC is acceptable only if tissue cannot be obtained for histological evaluation.
* ECOG Performance Status of 0 or 1
* Life expectancy of at least 12 weeks at the pre-treatment evaluation.
* Inoperable tumor (T2-T4, any N, M0 or M1 as defined by the TNM classification)
* Patient considered by the investigator to be appropriate for systemic therapy.
* Patients with at least one measurable lesion by CT-scan or MRI according to the Recist criteria, performed within 4 weeks prior to start of dosing.
* Patients who have not received any systemic anti-cancer treatment for HCC such as: chemotherapy, immunotherapy, hormonal therapy, vaccines as well as any systemic agent given with antineoplastic intent, prior to study inclusion. (previous local therapy is permitted). Previous treatment with Octreotide is however allowed, provided that the administration of the drug was discontinued at least 7 days prior enrolment or at least 28 days if the LAR (long acting release) formulation of the drug was used.
* Patients who have received local therapy, such as: surgery, radiation therapy, hepatic arterial embolization, chemo-embolization, radio-frequency ablation or cryo-ablation are eligible, provided that they either have a target lesion which has not been subjected to local therapy and/or the target lesion(s) within the field of the local therapy has shown an increase of 25% in the size. Furthermore, the local therapy applied to target or non-target lesions needs to have been completed at least 8 weeks prior to study inclusion (Lesions treated with external beam radiation therapy are not acceptable as target lesions, unless they fulfill the conditions described above).
* Adequate bone marrow, liver and renal function, as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin 8.5 g/dl
  * Absolute granulocytes 1.5 x 109/L
  * Platelet count 60 x 109/L
  * Total serum bilirubin 3 mg/dl
  * ALT (SGOT) and AST (SGPT) 5 x upper limit of normal
  * PT-INR 2.3 or PT 6 seconds above control
  * Serum creatinine 1.5 x upper limit of normal.
* Cirrhotic status of Child's Pugh class A or B. Child's Pugh class C should be excluded
* Written Informed Consent must be obtained and documented prior to any study specific procedures.

Exclusion Criteria:

Patients who meet the following criteria at the time of screening will be excluded; excluded medical conditions:

* Congestive heart failure defined as NYHA class III or IV.
* Serious cardiac arrhythmias.
* Active coronary artery disease or ischemia.
* Active clinically serious infections (> grade 2 NCI-CTC).
* Known history of HIV infection.
* Known metastatic brain or meningeal tumors.
* History of seizure disorder.
* History of organ allograft.
* Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis & T1] or other malignancies curatively treated > 3 years prior to entry).
* Patients with clinically significant gastrointestinal bleeding within the past month prior to study entry are ineligible.

Excluded therapies and medications, previous and concomitant:

* Any systemic anticancer treatment or any agent administered with antineoplastic intent, including chemotherapy, immunotherapy , vaccines or hormonal therapy given before study entry or during study treatment. Anticancer therapy is defined as any agent or combination of agents with clinically proven anticancer activity administered systemically, with the purpose of affecting the cancer, either directly or indirectly, including palliative and therapeutic endpoints. In certain cases, local anticancer therapy is allowed. See Inclusion Criteria for details.
* Any surgical procedure within 4 weeks prior to start of study drug.
* Autologous bone marrow transplant or stem cell rescue within 4 months of study entry.
* Use of biologic response modifiers, such as G-CSF, within 3 weeks of study entry. G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity, such as febrile neutropenia, when clinically indicated, or at the discretion of the investigator; however, they may not be substituted for a required dose reduction. Chronic Erythropoietin treatment prior to the study entry or during the study is permitted.
* Use of ritonavir and grapefruit juice.
* Prior use of Raf-Kinase inhibitors, MEK or Farnesyl Transferase Inhibitors. Any investigational drug therapy outside of this trial during or within 4 weeks of study entry.

Other Exclusion Criteria:

* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures (e.g. cervical cap, condom, diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between SORAFENIB and oral contraceptives.
* Substance abuse, medical, psychological or social conditions that, in the judgment of the investigator, is likely to interfere with the patient's participation in the study or evaluation of the study results.
* Known allergy to the investigational agent or any agent given in association with this trial.
* Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
N° of non progressive disease (complete and partial responses, stable disease) | 1 year

SECONDARY OUTCOMES:
Toxicity of the combination,ORR,Duration of responses, TTP and OS.PK, PD,Baseline pERK concentration, phospho VEGF-R2 concentration, plasma proteomics and gene expression profiling on blood cells and tumor biopsy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Oncologia, dei Trapianti e delle Nuove Tecnologie in Medicina ... Indirizzo: via Roma, 55 - 56100 Pisa Tel. 050-2218690 - Fax. 050-2218685, Pisa, Pisa, Italy

REFERENCES:
- [Derived] Petrini I, Lencioni M, Ricasoli M, Iannopollo M, Orlandini C, Oliveri F, Bartolozzi C, Ricci S. Phase II trial of sorafenib in combination with 5-fluorouracil infusion in advanced hepatocellular carcinoma. Cancer Chemother Pharmacol. 2012 Mar;69(3):773-80. doi: 10.1007/s00280-011-1753-2. Epub 2011 Oct 28. PMID 22033636